CLINICAL TRIAL: NCT06779994
Title: Safety and Efficacy of Streptococcus Salivarius Subsp. Thermophilus ST36 on Intestinal and Immune Function Improvement.
Brief Title: The Safety and Efficacy of Probiotic for Improving Intestinal and Immune Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wecare Probiotics Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: WK2025002
Record Dates: First submitted 2025-01-14; First posted 2025-01-17 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-08

CONDITIONS: Adults Aged 18-45 Years
MeSH Terms: interventions — Probiotics

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Double(Participant, investigator)
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Probiotic group (Experimental): 30B CFU/strip/day ST36, before meals; Storage: Store in a cool, dry place without sun exposure.
  Interventions: Dietary Supplement: Probiotic
- Placebo group (Placebo Comparator): Dextrin, one strip/day, before meals; Storage: Store in a cool, dry place without sun exposure.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Probiotic — The experimental phase of this study will last 8 weeks and each subject will have three visits (day 0, week 4 and week 8).
  Arms: Probiotic group
Dietary Supplement: Placebo — The experimental phase of this study will last 8 weeks and each subject will have three visits (day 0, week 4 and week 8).
  Arms: Placebo group

SUMMARY:
To evaluate the safety and efficacy of Streptococcus salivarius subsp. thermophilus ST36 in healthy adults on immune function and intestinal health.

ELIGIBILITY:
Inclusion Criteria:

* 1) Age 18-45 years; 2) Willing to undergo 3 follow-up visits during the intervention period; 3) Willing to provide 2 blood, urine, and stool samples during the intervention period; 4) Willing to self-administer Streptococcus salivarius subsp. thermophilus ST36/placebo once daily during the intervention period; 5) Good eyesight, able to read and write, and can wear glasses; 6) Have good hearing and be able to hear and understand all instructions during the intervention;

Exclusion Criteria:

* 1) Suffering from digestive disorders, mainly gastrointestinal disorders (celiac disease, ulcerative colitis, Crohn's disease); 2) Has a severe neurological condition (epilepsy, stroke, severe head trauma, meningitis within the past 10 years, brain surgery, brain tumor, prolonged coma - excluding general anesthesia); 3) Has received/is receiving treatment for the following psychiatric disorders: alcohol/drug/substance abuse dependence, schizophrenia, psychosis, bipolar disorder; 4) Take medication for depression or low mood; 5) Suffering from internal organ failure (heart, liver, or kidney failure, etc.); 6) Radiotherapy or chemotherapy in the past; 7) Surgery/procedure under general anesthesia within the past three years, or planned to undergo a procedure/procedure under general anesthesia within the next 3 months during this trial; 8) Have had hepatitis (hepatitis B, hepatitis C), HIV or syphilis in the past.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 98 (Actual)
Dates: Start 2025-04-10 (Actual); Primary Completion 2025-05-06 (Actual); Study Completion 2025-08-20 (Actual)

PRIMARY OUTCOMES:
Antimicrobial peptide levels in stool samples | 8 weeks
  Antimicrobial peptides refer to fecal calprotectin and LL-37(Cathelicidin Antimicrobial Peptide). The change in their concentrations at the end of the intervention was detected compared to baseline.

CONTACTS AND LOCATIONS:
Locations (1):
- Xu fei, Zhengzhou, Henan, China